CLINICAL TRIAL: NCT01816867
Title: Laparoscopic and Open Ventral Hernia Repair Using the Intramesh T1: a Prospective, Multicenter Registry
Brief Title: Laparoscopic and Open Ventral Hernia Repair Using the Intramesh T1
Status: Completed | Type: Observational
Sponsor: be Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BM-T1-08
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Ventral Hernia
Keywords: hernia; Treatment; laparoscopic; open technique
MeSH Terms: conditions — Hernia, Ventral; Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a ventral hernia
  Interventions: Device: Intramesh T1 implantation

INTERVENTIONS:
Device: Intramesh T1 implantation
  Other Names: Intramesh T1 Cousin Biotech

SUMMARY:
The purpose of the registry is to evaluate safety and efficacy of the Intramesh T1. This registry will collect data from 100 patients treated for a ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 18 years
* Written informed consent is obtained from patient
* Patient with a primary or incisional ventral hernia

Exclusion Criteria:

* Patient with a recurrent ventral hernia
* Patient with ASA class 5 and 6
* Patient underwent emergency surgery
* Patient is pregnant
* Patient with a known allergy to components of the ePTFE prosthesis
* Patient has a life expectancy less than 1 year
* Patient is unable to be compliant with the follow-up visits due to geographical, social or psychological factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a ventral hernia
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Recurrence rate at 12 months determined by clinical examination | 12 months

SECONDARY OUTCOMES:
Intraoperative complications | peri-procedural
  Defined as complications occurring during index-procedure from "skin-into-skin". The following events must be reported in the case report form:
  * enterotomy (bowel injury)
  * major bleeding requiring blood transfusion or reintervention
  * complications due to anesthesia
  * minor bleeding at a trocar insertion site
Post-operative complications | up to 30 days
  Defined as complications up to 30 days after index-procedure. The following events should be reported in the case report form:
  * local numbness
  * hematoma
  * seroma
  * superficial trocar site infection
  * mesh infection
  * hernia recurrence
  * death
Seroma | 1 month
  The rate of seroma at 1 month after index-procedure.
Freedom from hernia-related reinterventions | 12 months
  Reinterventions at 12 months after index-procedure
Late complications | 12 months
  Late complications at 12 months after index-procedure:
  * prolonged pain more than 8 weeks
  * local numbness
  * hernia recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Van der Speeten, MD, PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

REFERENCES:
- [Derived] Wen W, Majerus B, Van De Moortel M, Lobue S, Fobe D, Philippart P, Berwouts L, Coteur J, Gabriels K, Van der Speeten K. Laparoscopic ventral hernia repair using a composite mesh with polypropylene and expanded polytetrafluoroethylene: a prospective, multicentre registry. Acta Chir Belg. 2017 Oct;117(5):295-302. doi: 10.1080/00015458.2017.1313526. Epub 2017 Apr 25. PMID 28438090